CLINICAL TRIAL: NCT04452812
Title: Pilot Clinical, Statistical and Epidemiological Study on Efficacy and Safety of Convalescent Plasma for the Management of Patients With COVID-19
Brief Title: Statistical and Epidemiological Study Based on the Use of Convalescent Plasma for the Management of Patients With COVID-19
Acronym: PROMETEO
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Coahuila (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUS-001/2020
Record Dates: First submitted 2020-06-29; First posted 2020-06-30 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: COVID-19 Pneumonia; Convalescent Plasma
Keywords: COVID-19; Convalescent plasma; plasmapheresis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Pilot, experimental, randomized, prospective, longitudinal, clinical study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent plasma (Experimental): Best available treatment + convalescent plasma
  Best available treatment: hemodynamic support, oxygen supplementation, antibiotic therapy (if required), and individualized treatment judged by the attending physician.
  Plasma will be split by aliquots of 200 ml for its storage on -60 celsius degrees until it's used. After defrosting, it will be administered on 2 200 ml separated doses on a 12 hours interval.
  Interventions: Biological: Convalescent plasma
- Best available treatment (Placebo Comparator): Best available treatment + Placebo (0.9% saline solution)
  Best available treatment: hemodynamic support, oxygen supplementation, antibiotic therapy (if required), and individualized treatment judged by the attending physician.
  Placebo will consist on 2 doses of 200 ml of 0.9% saline solution separated on a 12 hour interval.
  Interventions: Biological: Convalescent plasma

INTERVENTIONS:
Biological: Convalescent plasma — Best available treatment + convalescent plasma
  Best available treatment: hemodynamic support, oxygen supplementation, antibiotic therapy (if required), and individualized treatment judged by the attending physician.
  Plasma will be split by aliquots of 200 ml for its storage on -60 celsius degrees until it's used. After defrosting, it will be administered on 2 200 ml separated doses on a 12 hours interval.

SUMMARY:
The health contingency established against the Severe Acute Respiratory Syndrome associated type 2 Coronavirus (SARS-CoV-2) has promoted a race against the clock for the search on treatment against the disease related with coronavirus (COVID-19). There are no current approved therapeutic options against the virus, although there is a rush for the development of drugs, vaccines and even the passive immunization through plasma from convalescent patients. This passive immunization is made with the administration of antibodies from patients that went through the infectious state of the disease and progress to clinical remission.

SARS-CoV-2, and its predecessor SARS-CoV-1, have great similarities between their genes and proteins; tis allow to hypothesize that the antibodies developed against SARS-CoV1 can recognize the antigens of SARS-CoV-2. In this manner, the transfusion of convalescent plasma to patients with the infection brings the probability on eliminating the infection, in this case SARS-CoV-2. There are evidence of this phenomenon observed in previous pandemics caused by SARS-CoV-1, Influenza AH1N1 and Ebola virus.

The objective of the study is to develop a therapeutic strategy based on the administration of plasma from patients with COVID-19 with clinical remission to patients that are coursing with the infection. The expected results hopes to establish an effective treatment and satisfactory recovery of patients with COVID-19. Also, we expect to describe the respective antibodies related against the SARS-CoV-2 infection.

DETAILED DESCRIPTION:
The health contingency established against the Severe Acute Respiratory Syndrome associated type 2 Coronavirus (SARS-CoV-2) has promoted a race against the clock for the search on treatment against the disease related with coronavirus (COVID-19). There are no current approved therapeutic options against the virus, although there is a rush for the development of drugs, vaccines and even the passive immunization through plasma from convalescent patients. This passive immunization is made with the administration of antibodies from patients that went through the infectious state of the disease and progress to clinical remission.

SARS-CoV-2, and its predecessor SARS-CoV-1, have great similarities between their genes and proteins; tis allow to hypothesize that the antibodies developed against SARS-CoV1 can recognize the antigens of SARS-CoV-2. In this manner, the transfusion of convalescent plasma to patients with the infection brings the probability on eliminating the infection, in this case SARS-CoV-2. There are evidence of this phenomenon observed in previous pandemics caused by SARS-CoV-1, Influenza AH1N1 and Ebola virus.

The objective of the study is to develop a therapeutic strategy based on the administration of plasma from patients with COVID-19 with clinical remission to patients that are coursing with the infection. The expected results hopes to establish an effective treatment and satisfactory recovery of patients with COVID-19. Also, we expect to describe the respective antibodies related against the SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria (Donors):

* Signed informed consent
* At least positive for 1 q-PCR test for SARS-CoV-2
* 14 days of COVID-19 clinical remission
* Positive serologic test for SARS-CoV-2
* Requirements to donate according to NOM-253-SSA1-2012
* To accept sample storing for future study

Inclusion Criteria (Receptors):

* Signed informed consent provided by the patient, legal guardian or the health provider if not available
* Patients hospitalized in an ICU dedicated to the treatment of COVID-19 patients
* At least positive for 1 q-PCR test for SARS-CoV-2
* Patients with COVID-19 defined as severe or critically ill:

Severe: RF > 30 bpm, oxygen saturation <94%, Pa/FiO2 <301, bilateral lung infiltrates that extends in >50% (by chest radiograph or CT scan) in 24-48 hours Critically ill: Respiratory failure (PaO2 <60 mmHg or SatO2 <90% with FiO2 >60%) and septic shock (MAP <65 mmHg with vasoactive requirement, lactate > 2 mmol/L and SOFA score >1)

Exclusion Criteria:

* Positive pregnancy test
* Patients in lactation
* Informed consent not signed
* Patients involved in other treatment protocols
* Patients on immunomodulatory drugs (DMARDs, monoclonal antibodies or smal molecule drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-07-06 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days
  Any cause mortality during the first 30 days of treatment
Side effects | 30 days
  Side effects associated with the administration of convalescent plasma

SECONDARY OUTCOMES:
Length of stay in Intensive Care Unit (ICU) | 14 days
  Time to discharge from the ICU
Length of stay in hospitalization | 21 days
  Time for discharge from hospital
Days of mechanical ventilation | 14 days
  Number of days with ventilatory support
Inflammatory biomarkers (d-dimer) | 21 days
  change in D-dimer (micrograms/L)
Inflammatory biomarkers (c-reactive protein) | 21 days
  change in C-reactive protein (milligrams/dL)
Inflammatory biomarkers (lactate dehydrogenase) | 21 days
  Change in LDH (UI/L)
Inflammatory biomarkers (ferritin) | 21 days
  Change in ferritin (nanograms/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario "Dr. Gonzalo Valdés Valdés", Saltillo, Coahuila, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol